CLINICAL TRIAL: NCT02114983
Title: Precision and Diagnostic Accuracy of General Practitioner-performed Compression Ultrasound for Proximal Symptomatic Deep Vein Thrombosis
Brief Title: General Practitioner-performed Compression Ultrasound for Deep Vein Thrombosis
Status: Completed | Type: Observational
Sponsor: Azienda Sanitaria Locale ASL 6, Livorno (Other Government)
Responsible Party: Principal Investigator, Nicola Mumoli, Dr Nicola Mumoli, M.D., Azienda Sanitaria Locale ASL 6, Livorno
Other Study IDs: MN-1
Record Dates: First submitted 2014-04-13; First posted 2014-04-15 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Deep Vein Thrombosis
Keywords: deep vein thrombosis; diagnostic accuracy; general practitioner; test; compression ultrasonography; ultrasound
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: d-dimer
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- first episode of suspected DVT of the lower limbs: patients with first suspected episode of DVT of the lower limbs
  Interventions: Other: compression ultrasonography

INTERVENTIONS:
Other: compression ultrasonography — CUS in patients with a high pre-test clinical probability of DVT and/or a positive D-dimer

SUMMARY:
Numerous studies have demonstrated excellent diagnostic accuracy of Compression Ultrasonography (CUS) performed by hospitals doctors, skilled and unskilled in Radiology.

Recently, it was demonstrated that adequately ultrasonography-trained General Practitioners (GP) can perform reliable ultrasound to increase the speed and improve the quality of clinical management of various clinical conditions. To date, in the medical literature there are no studies that demonstrate the diagnostic accuracy of GP in performing CUS for the diagnosis of Deep Vein Thrombosis (DVT). Therefore, we plan to perform a prospective, multicenter, cohort study in which a large number of consecutive outpatients with symptoms or signs of DVT are subject to the CUS by the GP with the aim of evaluating the precision and the diagnostic accuracy compared to specialists in vascular ultrasound, which in this case will be the standard of reference.

ELIGIBILITY:
Inclusion Criteria:

* first episode of DVT of lower limbs

Exclusion Criteria:

* previous episodes of DVT
* ongoing anticoagulation
* age younger than 18 years
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All outpatients evaluated at home or at office by the GP with a first episode of suspected DVT of the lower limbs will be screened with CUS. GP may use his/her own ultrasound, or take advantage of the equipment of the Vascular Service of the Hospital. Shortly afterward, (i.e., within 2 hours), all outpatients will be re-evaluated by a doctor with expertize in vascular ultrasound
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of General Practitioner in performing CUS for the diagnosis of DVT | Up to 2 h hours after ambulatory admission
  Aim of our study is to perform a prospective, multicenter, cohort study in which a large number of consecutive outpatients with symptoms or signs of DVT are subject to the CUS by the General Practitioner with the aim of evaluating the diagnostic accuracy.

SECONDARY OUTCOMES:
Precision of CUS performed by General Practitioner for the diagnosis of DVT | Up to 2 h hours after ambulatory admission
  The secondary outcome of the study will be the the precision of CUS performed by a doctor of general medicine for the diagnosis of proximal DVT of the lower limbs with respect to the medical specialist in vascular diagnostics, in this case used as a reference.

OTHER OUTCOMES:
To assess the prevalence of DVT in patients with a high pre-test probability and/or a positive D-dimer | Up to 2 h hours after ambulatory admission

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Mumoli, MD, Principal Investigator — Section of Vascular Medicine - Livorno Hospital, Italy
Locations (1):
- Azienda USL 6 Livorno, Livorno, Tuscany, Italy